CLINICAL TRIAL: NCT04426682
Title: In Patients Who Underwent Incontinence Surgery and Who Had Postoperative Recurrence Comparison of Urodynamics Parameters Performed in Preoperative and Postoperative Period
Brief Title: Incontinence Surgery and Urodynamics Parameters
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Pınar Kadiroğulları M.D, Department of Obstetrics and Gynecology,Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: ATADEK / 2020.06
Record Dates: First submitted 2020-06-05; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Incontinence; Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post-operative urinary incontinents: In patients who have previously had incontinence surgery due to stress incontinence, symptoms may return in the following years, and the patient may reapply with urinary incontinence. The first group will consist of postoperative urinary incontinence recurrent patients. Patients whose urodynamics are reperformed due to recurrence are the study group.
  Interventions: Diagnostic Test: urodynamics parameters
- without postoperative urinary incontinence: Patients who previously had incontinence surgery due to stress incontinence and who did not have postopertive urinary incontinence but whose urodynamics were repeated during the routine controls will constitute the control group.
  Interventions: Diagnostic Test: urodynamics parameters

INTERVENTIONS:
Diagnostic Test: urodynamics parameters — Urodynamics evaluation is performed in the preoperative period in patients whose operation is planned due to incontinence.
  Urodynamics evaluation is performed again in patients who applied with postoperative relapse due to surgery failure or different reasons.
  It will be shown whether there is a difference between the urodynamics parameters of preoperatively examined patients and those of urodynamics examined in case of postoperative failure.

SUMMARY:
In patients who have previously had incontinence surgery due to stress incontinence (Midurethral slings (tvt, tot, etc.)), the symptoms may return in the following years and the patient can reapply with urinary incontinence. Urodynamic evaluation is important before stress incontinence surgery to confirm clinical diagnosis based on symptoms and findings and to determine the factors that may affect the effectiveness of surgery and the possibility of complications. Urodynamics evaluation is performed in the preoperative period in patients scheduled for incontinence. Urodynamics evaluation is performed again in patients who applied with post-operative recurrence due to surgery failure or different reasons.

It is aimed to show whether there is a difference between the urodynamics parameters of these patients who were examined preoperatively and the urodynamics parameters examined in case of postoperative failure. Thus, the primary goal; to show which of these parameters has deterioration or if the surgical method is insufficient if it is within certain limits or urinary incontinence may recur.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously undergone surgery for stress incontinence
* Those who are symptomatic again in their post-operative follow-up (urinary incontinence),
* Patients who underwent preoperative and postoperative urodynamics

Exclusion Criteria:

* Those with chronic diseases or medications that may cause urinary incontinence
* Patients with mixed or urge incontinence
* Patients who are not symptomatic postoperatively

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The files of the patients will be accessed through the system, and patients who have had incontinence surgery and applied again due to recurrence will be selected. The data of these patients will be scanned and recorded. The control group will also be created in the same way, and data of patients who have undergone surgery and have no urinary incontinence and who have postoperative urodynamics will be recorded. .
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
urodynamics parameters V max | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; V max (voiding speed) cm3
urodynamics parameters bladder complians | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; bladder complians
urodynamics parameters valsalva leak point pressure | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; valsalva leak point pressure (mmhg)
urodynamics parameters abdominal leak point pressure | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; abdominal leak point pressure (mmhg)
urodynamics parameters P det | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; P detrusitor (P det) (mmhg)
urodynamics parameters P abd | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; P abdominal (P abd) (mmhg)
urodynamics parameters P urethral | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; P urethral (mmhg)
urodynamics parameters UPP | 5 YEARS
  urodynamics parameters of patients before and after surgery will be examined urodynamic parameters to look at; urethral pressure profile (UPP)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)